CLINICAL TRIAL: NCT02132338
Title: Evaluation of the Educational Program of Diabetes Mellitus: Focus on Empowerment
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, HELOISA DE CARVALHO TORRES, Postdoctoral, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CAAE 22372013.2.000.5149
Record Dates: First submitted 2014-04-22; First posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Prevention; Health Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The Education Health Program (Experimental): Intervention forth knowledge and attitudes necessary for self-care
  Interventions: Behavioral: The Education Health Program

INTERVENTIONS:
Behavioral: The Education Health Program — The operation of the educational program for the group under intervention will consist of groups operating with the triad of diabetes mellitus (pathophysiology of the disease, physical activity and diet), to be held in five times (cycles) approach, an interval of three months being held between them . In each session, participants will be the same (under multidisciplinary team intervention), the content will also be the same, however, using different educational strategies. During the intervals between cycles these users will be monitored by phone by equity and / or nursing students of the Federal University of São João Del Rei properly trained to do so. The educational program will be developed in five times (T0, T3, T6, T9, T12) and with an interval of three months. At every moment the educational process will be conducted with three consecutive meetings with one week interval. In summary, 15 educational sessions with the experimental group will be held.
  Other Names: Provide knowledge;; Attitudes;; and skills to care self-management and empowerment of diabetes mellitus.

SUMMARY:
With health education, patients will have knowledge of the disease and may modify their attitudes to diabetes. Have a different behavior, will perform self-management of their health. Will adhere to physical activity, the better control of the disease and have quality of life. Empower the patient through the educational practices.

DETAILED DESCRIPTION:
In this sense, from the perspective that the routine monitoring of users with type 2 diabetes should be performed at the primary health care, which has the structural axis the family health team, and that education is fundamental to the self-management of diabetes mellitus care, applying a evaluative research based on an educational program to check before and after clinical, anthropometric data and validated instruments can provide an effective means of control and prevention of disease.

The purpose of randomization is to compare the effects and values of the dependent variables ( knowledge about diabetes mellitus, psychological attitudes, adherence to practices related to physical activity and diet self-care, empowerment for self-care in diabetes mellitus and control of clinical indicators ) in the experimental group with the group control, which are associated with the independent variable ( educational program). For the experimental group an educational systematized process, to evaluate the scope for enhancing the educational process with emphasis on Diabetes empowerment to provide self-care, thereby improving disease control will be performed. Have the control group will maintain the traditional care through individual consultations and information about the disease, through leaflets that could assist in the educational process for self-management of care. All subjects in the experimental group and the control group will be questioned in the pre -test and post - test by related instruments: (1) knowledge of the diabetes mellitus, (2) attitudes toward the psychological aspects, (3) self-care (medication adherence, diet and physical activity), (4) empowerment for self-care in diabetes mellitus and (5) clinical indicators.

ELIGIBILITY:
Inclusion Criteria:

* users from 30 years of age diagnosed with type 2 diabetes mellitus,
* degree of education above the fourth grade of elementary education and
* ability to attend the education program.

Exclusion Criteria:

* users with reading disability and
* chronic complications (defined as kidney failure, blindness, amputation of limbs, etc.).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin level before and after intervention | 1 year after start of the intervention
  The intervention groups will be followed for 1 year. During this period glycated hemoglobins in time 0,3,6 and 12 months will be harvested.

SECONDARY OUTCOMES:
level of knowledge about diabetes mellitus | 1 year after start of the intervention
  The intervention and control groups will be followed for 1 year. During this period glycated hemoglobins in time 0,3,6 and 12 months will be harvested.
diabetes mellitus empowerment for self-care | 1 year after start of the intervention
  The intervention and control groups will be followed for 1 year. During this period glycated hemoglobins in time 0,3,6 and 12 months will be harvested.
tests such as cholesterol | 1 year after start of the intervention
  The intervention and control groups will be followed for 1 year. During this period glycated hemoglobins in time 0,3,6 and 12 months will be harvested.
tests such as fasting glucose | 1 year after start of the intervention
  The intervention and control groups will be followed for 1 year. During this period glycated hemoglobins in time 0,3,6 and 12 months will be harvested.
body mass index | 1 year after start of the intervention
  The intervention and control groups will be followed for 1 year. During this period glycated hemoglobins in time 0,3,6 and 12 months will be harvested.

OTHER OUTCOMES:
Loss of participants in the intervention by forfeit | 1 year after start of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Heloisa Carvalho Torres, posdoctor, Study Director — Federal University of Minas Gerais; Daniel Nogueira Cortez, master, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Derived] Cortez DN, Macedo MM, Souza DA, Dos Santos JC, Afonso GS, Reis IA, Torres HC. Evaluating the effectiveness of an empowerment program for self-care in type 2 diabetes: a cluster randomized trial. BMC Public Health. 2017 Jan 6;17(1):41. doi: 10.1186/s12889-016-3937-5. PMID 28061840